CLINICAL TRIAL: NCT06807294
Title: Feasibility Testing of a Tai Chi Program for Chemotherapy-Induced Peripheral Neuropathy Treatment (TCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ting Bao, MD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-399
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN); Peripheral Neuropathy Due to Chemotherapy; Peripheral Neuropathies; Neuropathy
Keywords: Peripheral Neuropathy; Chemotherapy Induced Peripheral Neuropathy; Cancer survivor; CIPN; Tai Chi; Balance training; Falls prevention; Non-pharmacological intervention; Mind-body exercise; Quality of life; Feasibility study; Pilot study
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Tai Chi Treatment Group (Experimental): 14 randomized participants will complete:
  * 1 baseline visit session.
  * Virtual Tai Chi session 2x weekly (60 minutes per session).
  * Independent Tai Chi sessions 3 days a week (60 minutes per session).
  * 12 week follow up visit.
  Interventions: Behavioral: Tai Chi Program
- Arm B: Waitlist Control Group (No Intervention): 7 randomized participants will complete:
  * 1 baseline visit session
  * Standard CIPN care prescribed by primary care physician/oncologist.
  * 12 week follow up visit
  * Participants will be offered 24 complimentary, virtual, Tai Chi training sessions over 12 weeks after completion of the 12-week follow-up visit.

INTERVENTIONS:
Behavioral: Tai Chi Program — 12-week virtual Tai Chi program with experienced Tai Chi instructor. Sessions will be conducted via the HIPPA-compliant teleconference platform, Zoom.
  Arms: Arm A: Tai Chi Treatment Group

SUMMARY:
This research is being done to determine whether a 12-week virtual Tai Chi training program, designed to improve balance and small nerve fiber function, is feasible and acceptable among cancer survivors with chemotherapy-induced peripheral neuropathy (CIPN).

DETAILED DESCRIPTION:
This is a prospective, randomized, waitlist-controlled pilot trial to examine the suitability of the virtual Tai Chi program in cancer survivors with CIPN. Tai Chi is a mind-body practice that involves gentle body movements, meditation, and breathing techniques. It has proven to be effective in enhancing balance control and relieving musculoskeletal pains.

This study randomly assigns cancer survivors with CIPN with self-perceived balance difficulties to one of two groups: Group A Tai Chi Group versus Group B Waitlist Group. Randomization means a participant is placed into a study group by chance.

The research study procedures including screening for eligibility, questionnaires, and sensory and functional testing.

Participation in this study is expected to last for up to 12 weeks.

It is expected that about 21 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and older
* Cancer survivors with no evidence of disease (cancer);
* Completed neurotoxic chemotherapy, i.e., platinum agents, taxanes, vinca alkaloids, and bortezomib, at least three months before enrollment;
* A CIPN diagnosis based on symptom history, loss of deep tendon reflexes, or presence of symmetrical stocking-glove pain, numbness, or paresthesia;
* Answers "yes" to the following question: "Do you feel as though your balance is affected from experiencing CIPN?" or "Are you afraid of falling as a result of your CIPN?";
* On a stable regimen (no change in past three months) if taking anti-neuropathy or other pain medications;
* Eastern Cooperative Oncology Group (ECOG) Performance Status Scale score ≤ 2
* Willing to adhere to all study-related procedures, including randomization to the Tai Chi or waitlist group, 2 in-person visits to Dana-Farber Cancer Institute (DFCI) (one within 2 weeks of enrollment and one at week 12);
* Willing to adhere to requirement that no new pain medication be taken throughout the study period; and
* Individuals receiving endocrine therapy or targeted/antibody therapy, such as trastuzumab, pertuzumab, or immunotherapy, will be eligible to participate.

Exclusion Criteria:

• Patients who have received physical therapy or Tai Chi training, specifically for CIPN, in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate for the Tai Chi Program | 6 months
  The intervention is considered feasible if 21 participants are enrolled within the first 6 months of the study period.
Assessment Completion Rate | 12 weeks
  The intervention is considered feasible if 75% of all evaluable participants, 16 out of 21, complete the biobehavioral assessments during the intervention period.
Session Completion Rate | 12 weeks
  The intervention is considered feasible if 62% of participants in the intervention arm, 9 out of 14, attend at least 80% or 20 of the 24 online sessions.
Acceptability of Intervention Measure (AIM) Score | 12 weeks
  Assessed by the Acceptability of the Intervention Measure (AIM), a 4-item measure rated on a 5-point Likert scale with answers ranging from "Completely disagree" to "Completely agree." A total scores range is 4 to 20 with a higher score indicating greater acceptability.

SECONDARY OUTCOMES:
Consent Rate (Arm A) | Up to 6 months (based on total accrual duration)
  Defined as the proportion of participants enrolled out of those eligible for study entry.
Consent Rate (Arm B) | Up to 6 months (based on total accrual duration)
  Defined as the proportion of participants enrolled out of those eligible for study entry.
Change in balance, strength, gait health and mobility factors from Baseline to 12 Weeks (Arm A) | Baseline and 12 weeks
  Assessed by the Berg Balance Scale (BBS), the incidence of falls, fall-related injuries, the Functional Reach Test (FRT) to measure dynamic balance and muscle flexibility (lower scores indicating higher fall risk), the Single Leg Stance Test (SLS) to evaluate static balance with eyes open and closed (abnormal values indicating balance impairment), the Timed Up and Go (TUG) test, the 30-second Chair Stand (30CS) test to assess motor performance (with lower TUG scores and higher 30CS scores reflecting better functional balance, strength, and endurance), and gait speed measurement across an 8-meter hallway under three conditions (quiet walking, fast speed, and cognitive dual task) at baseline and after 12 weeks of Tai Chi training.
Change in balance, strength, gait health and mobility factors from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  Assessed by the Berg Balance Scale (BBS), the incidence of falls, fall-related injuries, the Functional Reach Test (FRT) to measure dynamic balance and muscle flexibility (lower scores indicating higher fall risk), the Single Leg Stance Test (SLS) to evaluate static balance with eyes open and closed (abnormal values indicating balance impairment), the Timed Up and Go (TUG) test, the 30-second Chair Stand (30CS) test to assess motor performance (with lower TUG scores and higher 30CS scores reflecting better functional balance, strength, and endurance), and gait speed measurement across an 8-meter hallway under three conditions (quiet walking, fast speed, and cognitive dual task) at baseline and after 12 weeks of Tai Chi training.
Change in Berg Balance Scale (BBS) Score from Baseline to 12 Weeks (Arm A) | Baseline and 12 weeks
  Assessed by the BBS, a 14-item tool to measure participant balance ability. Each task is scored on a scale from 0 to 4 with a total scores range of 0 to 56. A higher score indicates better balance.
Change in Berg Balance Scale (BBS) Score from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  Assessed by the BBS, a 14-item tool to measure participant balance ability. Each task is scored on a scale from 0 to 4 with a total scores range of 0 to 56. A higher score indicates better balance.
Change in Fall Rate from Baseline to 12 Weeks (Arm A) | Baseline and 12 weeks
  Defined as the number of falls which occur during the intervention period. A fall is an unplanned descent to the floor with or without injury according to the National Database of Nursing Quality Indicators (NDNQI) definition. Falls included are 1) those occurring on a surface where caregivers and clinicians do not expect to find a participant, and 2) falls unassisted or assisted, and 3) falls from rolling off a low bed.
Change in Fall Rate from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  Defined as the number of falls which occurred during the intervention period. A fall is an unplanned descent to the floor with or without injury according to the National Database of Nursing Quality Indicators (NDNQI) definition. Falls included are 1) those occurring on a surface where caregivers and clinicians do not expect to find a participant, and 2) falls unassisted or assisted, and 3) falls from rolling off a low bed.
Change in the Number of Fall-Related Injuries from Baseline to 12 Weeks (Arm A) | Baseline and 12 weeks
  As defined by the NDNQI definitions for fall-related injuries. Injuries will be recorded by the participant in the supplied home diary and will be summarized descriptively.
Change in the Number of Fall-Related Injuries from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  As defined by the NDNQI definitions for fall-related injuries. Injuries will be recorded by the participant in the supplied home diary and will be summarized descriptively.
Change in Timed-Up-And-Go (TUG) Test from Baseline to 12 Weeks (Arm A) | Baseline to 12 weeks
  Assessed by the TUG Test. Participants are instructed to stand up from a chair, walk three meters as quickly and safely as possible, turn around, walk back, and sit down. The test is timed in seconds, with a longer time indicating worse performance. Nine seconds is the cutoff for high risk of falls.
Change in TUG Test from Baseline to 12 Weeks (Arm B) | Baseline to 12 weeks
  Assessed by the TUG Test. Participants are instructed to stand up from a chair, walk three meters as quickly and safely as possible, turn around, walk back, and sit down. The test is timed in seconds, with a longer time indicating worse performance. Nine seconds is the cutoff for high risk of falls.
Change in Brief Pain Inventory-Short For (BPI-SF) Score from Baseline to 12 Weeks (Arm A) | Baseline to 12 weeks
  Assessed by the BPI-SF, 9-item measure of the severity of pain and pain interference in the 24 hours prior to questionnaire administrations. A simple numeric rating scale from 0 to 10 is used for item rating, and a total score is the mean of the item ratings. Higher scores indicate greater pain intensity and greater interference with function.
Change in BPI-SF Score from Baseline to 12 Weeks (Arm B) | Baseline to 12 weeks
  Assessed by the BPI-SF, 9-item measure of the severity of pain and pain interference in the 24 hours prior to questionnaire administrations. A simple numeric rating scale from 0 to 10 is used for item rating, and a total score is the mean of the item ratings. Higher scores indicate greater pain intensity and greater interference with function.
Change in the Neurotoxicity (Ntx) Subscale Score from Baseline to 12 Weeks (Arm A) | Baseline to 12 weeks
  Assessed by the Ntx Subscale of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG) questionnaire. The Ntx Subscale is an 11-item measure of symptoms in the 7 days prior to questionnaire administration. Answers are rated on a 5-point Likert scale ranging from 0 "Not at all" to 4 "Very much" with a total scores range of 0 to 44. Higher scores represent higher functioning and fewer or less severe CIPN symptoms.
Change in the Neurotoxicity (Ntx) Subscale Score from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  Assessed by the Ntx Subscale of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG) questionnaire. The Ntx Subscale is an 11-item measure of symptoms in the 7 days prior to questionnaire administration. Answers are rated on a 5-point Likert scale ranging from 0 "Not at all" to 4 "Very much" with a total scores range of 0 to 44. Higher scores represent higher functioning and fewer or less severe CIPN symptoms.
Change in Tactile Threshold Value from Baseline to 12 Weeks (Arm A) | Baseline and 12 weeks
  This will be measured using a set of 20 Von Frey monofilaments. With participant's eyes closed, and starting at the smallest size filament, the clinical research coordinator (CRC) will touch the testing site at a 90-degree angle to the site surface until the filament bends for a one second duration. The CRC will continue this with ascending filament size in order until the participant reports feeling a touch sensation at the testing location. The force at which touch is perceived will be recorded as the tactile threshold. Tactile threshold will be assessed at the dorsum of the interphalangeal joint of the right and left big toes. Value will be recorded as the average of three readings.
Change in Tactile Threshold Value from Baseline to 12 Weeks (Arm B) | Baseline and 12 weeks
  This will be measured using a set of 20 Von Frey monofilaments. With participant's eyes closed, and starting at the smallest size filament, the clinical research coordinator (CRC) will touch the testing site at a 90-degree angle to the site surface until the filament bends for a one second duration. The CRC will continue this with ascending filament size in order until the participant reports feeling a touch sensation at the testing location. The force at which touch is perceived will be recorded as the tactile threshold. Tactile threshold will be assessed at the dorsum of the interphalangeal joint of the right and left big toes. Value will be recorded as the average of three readings.
Change in Vibration Threshold Value from Baseline to 12 weeks (Arm A) | Baseline to 12 weeks
  This will be assessed using a handheld biothesiometer and the amplitude of vibration will be gradually increased (1 volt/second) until the sensation of vibration is first perceived by the participant. The average of three perception thresholds at the dorsal interphalangeal joint of the dominant big toe will be recorded as the vibration threshold.
Change in Vibration Threshold Value from Baseline to 12 weeks (Arm B) | Baseline to 12 weeks
  This will be assessed using a handheld biothesiometer and the amplitude of vibration will be gradually increased (1 volt/second) until the sensation of vibration is first perceived by the participant. The average of three perception thresholds at the dorsal interphalangeal joint of the dominant big toe will be recorded as the vibration threshold.
Change in the Short Falls Efficacy Scale - International (Short FES-I) from Baseline to 12 Weeks (Arm A) | Baseline to 12 weeks
  Assessed by the Short FES-I, a 7-item measure of concerns about falls during daily activities. Answers are rated on a 4-point scale ranging from 1 "Not at all concerned" to 4 "Very concerned" with a total scores range of 7 to 28. A higher score represents greater participant concern.
Change in the Short Falls Efficacy Scale - International (Short FES-I) from Baseline to 12 Weeks (Arm B) | Baseline to 12 weeks
  Assessed by the Short FES-I, a 7-item measure of concerns about falls during daily activities. Answers are rated on a 4-point scale ranging from 1 "Not at all concerned" to 4 "Very concerned" with a total scores range of 7 to 28. A higher score represents greater participant concern.
Change in Functional Reach Test from Baseline to 12 Weeks (Arm A) | Baseline to 12 weeks
  The FRT test is used to quantify balance ability. A participant is instructed to flex the test arm forward to 90 degrees and to reach forward as far as possible before taking a step. The reach is determined by the total excursion of the third metacarpal from the starting point (with the handheld in a fist) to the point just before balance is lost. The final score is the average of three measurements.
Change in Functional Reach Test from Baseline to 12 Weeks (Arm B) | Baseline to 12 weeks
  The FRT test is used to quantify balance ability. A participant is instructed to flex the test arm forward to 90 degrees and to reach forward as far as possible before taking a step. The reach is determined by the total excursion of the third metacarpal from the starting point (with the handheld in a fist) to the point just before balance is lost. The final score is the average of three measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- See also: Recruitment Website — https://rally.massgeneralbrigham.org/study/tctstudy